CLINICAL TRIAL: NCT01036165
Title: A Twelve-week, Phase IIIb, Open-label, Single-arm, Multicenter Trial to Evaluate Ease of Use of an Electronic Autoinjector (RebiSmart™) for Self-injection in Subjects With Relapsing Multiple Sclerosis (RMS) Treated With Rebif® 44mcg Subcutaneously (sc) Three Times a Week (Tiw)
Brief Title: A Multicenter, Open-label, RebiSmart™ Autoinjector Ease of Use Study
Acronym: Performs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Responsible Party: Ahmad Al-Sabbagh, Vice President Medical Affairs Neurology, EMD Serono, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 29652
Record Dates: First submitted 2009-12-18; First posted 2009-12-21 (Estimated); Results first posted 2010-12-22 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: RebiSmart™ — The RebiSmart™ autoinjector contains Rebif® 132 mcg multidose cartridges for sc injection.

SUMMARY:
The purpose of this study is to test the RebiSmart™ for

* ease of use
* multiple domains related to subject's acceptability and satisfaction
* reliability of the correct function for self-injection of Rebif® 44 mcg sc tiw in subjects with RMS.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects, 18-65 years of age, inclusive, at the time of informed consent signature
2. RMS diagnosed according to the McDonald criteria
3. Currently receiving Rebif® 44mcg sc tiw using manual injections and/or Rebiject II autoinjector for greater than or equal to twelve weeks
4. Capable of self-injecting using the RebiSmart™ autoinjector. Self- injecting is defined as being able to make 2 of the 3 weekly injections without assistance.
5. Be willing and able to comply with the study procedures for the duration of the trial
6. Have given written informed consent and signed Health Insurance Portability and Accountability Act (HIPAA) Authorization before any study- related activities are carried out
7. Female subjects must not be either pregnant or breast-feeding and must lack childbearing potential, as defined by either:

   * Being post-menopausal or surgically sterile, or using a highly effective method of contraception (defined as a method that results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly, and includes for instance, implants, injectables, combined oral contraceptives*, some intrauterine devices, sexual abstinence or vasectomised partner)
   * Female subjects of childbearing potential must have a negative pregnancy test at Screening and Study Day 1 to be included in the trial. A urine pregnancy test will also be done at the Week 12/Exit visit

     * Note for subjects using a hormonal contraceptive method: No formal drug interaction studies have been carried out with Rebif®. As interferons have been reported to exert an inhibitory activity on hepatic microsomal enzymes, it is unlikely that the clearance of oral contraceptives would increase and result in decreased efficacy. In over 10,000 patient years of clinical trial experience with Rebif®, there has never been any indication of an interaction with oral contraceptives.

Exclusion Criteria:

1. Have used any other injectable medications (e.g. for pain) on a regular basis during the week prior to Screening or throughout the duration of the trial (the administration of a single injection for treatment or prophylaxis of a condition unrelated to MS or Rebif® therapy (e.g., influenza or pneumococcus vaccination) will be acceptable)
2. Have received MS therapy other than Rebif® within twelve weeks prior to Screening or at any time during the trial (e.g., other disease modifying drugs, Rebif® New Formulation, combination therapy, immunomodulatory and/or immunosuppressive agents, including but not limited to any other interferon (Avonex/Betaseron/Extavia), glatiramer acetate (Copolymer I), cyclophosphamide, cyclosporine, methotrexate, linomide, azathioprine, mitoxantrone, teriflunomide, laquinimod, cladribine, fingolimod (FTY720), total lymphoid irradiation, anti-lymphocyte monoclonal antibody treatment (e.g. natalizumab, alemtuzumab/Campath, anti-CD4), Intravenous immunoglobulin (IVIg), cytokines or anti-cytokine therapy) and telbivudine
3. Have inadequate liver function, defined by a alanine aminotransferase (ALT) > 2.5x upper limit of normal (ULN), or alkaline phosphatase > 2.5x ULN, or total bilirubin > 2.5x ULN
4. Have inadequate bone marrow reserve, defined as a total white blood cell count < 3.0x 109/L, platelet count < 75x109/L, hemoglobin < 100g/L
5. Have complete transverse myelitis or simultaneous-onset bilateral optic neuritis
6. Have a history of alcohol or drug abuse
7. Have thyroid dysfunction
8. Have moderate to severe renal impairment
9. Have a major medical or psychiatric illness that in the opinion of the investigator creates undue risk to the subject or could affect compliance with the study protocol
10. Have a history of seizures not adequately controlled by treatment
11. Have serious or acute cardiac disease, such as uncontrolled dysrhythmias, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure
12. Have, in the opinion of the investigator, major visual, physical or cognitive impairment that would preclude the subject from self-injecting with the RebiSmart™ autoinjector
13. Have a known hypersensitivity or allergy to interferon-beta or any of the excipients
14. Have participated in another clinical trial within the past thirty days
15. Are pregnant or attempting to conceive
16. Have previously used a RebiSmart™ autoinjector

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2010-01; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dangond, MD, Study Director — EMD Serono
Locations (1):
- EMD Serono, Inc., Rockland, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 103 subjects were recruited from 15 US clinics in the US during the trial period February 2010 to August 2010
Pre-assignment Details: Subjects who signed informed consent and satisfied the eligibility critera at screening returned to the clinic on study day 1 to begin treatment with the Rebismart autoinjector. All subjects participating in the trial received Rebif 44 mcg sc tiw using the Rebismart autoinjector for 12 weeks.
Groups:
- Subject Disposition: Intent-to-Treat Analysis
Period: Overall Study
Arm/Group | Subject Disposition
Started | 103
Completed | 88
Not Completed | 15
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 3
Not completed — Device Related Issues | 3
Not completed — Problems finding proper area to inject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subject Disposition
Number analyzed (Participants) | 103
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 103
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.4 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 103

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint is the Proportion of RMS Subjects Rating the RebiSmart™ Autoinjector as 'Easy to Use' or 'Very Easy to Use' for Self-injection in a User Trial Questionnaire.
Description: Data from the User Trial Questionnaire-B, Question 13 (Overall, how do you rate your experience with using the injection device). Mean and confidence intervals refer to proportion of subjects responding positively to question. Missing values were replaced with worst case response.
Time Frame: at 12 Weeks
Measure: Mean (95% Confidence Interval); unit: Proportion of subjects
Arm/Group | Subject Disposition
Number analyzed (Participants) | 103
Proportion of subjects | 0.78 [0.70 to 0.86]
Statistical Analysis 1: Comparison: Subject Disposition; Test type: Superiority or Other; Mean positive response = 0.78, 95% CI 2-sided [0.70 to 0.86] — Confidence Interval calculated from normal approximation to the binomial. The primary objective was met if the lower limit of the 95% confidence interval was >0.50

2. Secondary Outcome: Multiple Secondary Endpoints Will be Assessed, Based on Questions From the User Trial Questionnaire Related to the RebiSmart™ Autoinjector Use-related Outcomes.
Description: The User Trial Questionnaire B was administered at Week 6 and Week 12 to assess the ease of use, functional reliability, overall satisfaction, satisfaction with device attributes, convenience, safety and portability of the Rebismart. Means and confidence intervals refer to the proportion of subjects responding positively, based on the number of non-missing values for each question. Secondary endpoints presented for decriptive purposes only thus no statistical analysis performed.
Time Frame: at Week 12
Measure: Mean (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Subject Disposition
Number analyzed (Participants) | 103
Percentage of subjects
  Device makes injections simple | 81.8 [73.8 to 89.9]
  Allows easy access to skin injection sites | 79.5 [71.1 to 88.0]
  Helps me self-administer Injections | 84.1 [76.4 to 91.7]
  Step by step Instructions are a key benefit | 93.2 [87.9 to 98.4]
  Ease of using injection device | 90.9 [84.9 to 96.9]
  Ease of loading cartridge | 97.7 [94.6 to 100.0]
  Ease of inserting the needle | 84.1 [76.4 to 91.7]
  Ease of pushing the button | 96.6 [92.8 to 100.0]
  Ease of holding device during injection | 84.1 [76.4 to 91.7]
  Ease of removing the needle from device | 76.1 [67.2 to 85.0]
  Able to often or always administer full injection | 98.9 [96.6 to 100.0]
  Rate the convenience of the device | 87.5 [80.6 to 94.4]

ADVERSE EVENTS:
Arm/Group | Subject Disposition
Serious Adverse Events (participants affected / at risk) | 1/99
Other Adverse Events (participants affected / at risk) | 92/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject Disposition (N=99)
Appendicitis (Infections and infestations) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subject Disposition (N=103)
Influenza like illness (General disorders) | 11 (11)
Injection site erythema (General disorders) | 35 (35)
Injection site haematoma (General disorders) | 12 (12)
Injection Site Pain (General disorders) | 52 (52)
Urinary Tract Infection (General disorders) | 8 (8)
Headache (Nervous system disorders) | 6 (6)
Multiple Sclerosis relapse (Nervous system disorders) | 9 (9)
Injection site haemorrhage (General disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Neither Institution nor any Principal Investigators shall publish or present any results from such Study to any third parties until: (i) EMD Serono publishes the results from all sites participating in such Study; (ii) Institution receives notification from EMD Serono that publication of the multi-site results is no longer planned; or (iii) twenty-four (24) months following the completion of the multi-site study at all sites, whichever occurs first.